CLINICAL TRIAL: NCT04004858
Title: Reducing Acute Rectal Toxicity for Hypofractionated Prostate Radiotherapy - An Multi-institution Pilot Study of Reduced PTV Margin
Brief Title: Prostate Margin Reduction to Reduce Acute Rectal Toxicity (PROTRACT)
Acronym: PROTRACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southlake Regional Health Centre (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Beibei Zhang, Medical Physicist, Southlake Regional Health Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 043-1819
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: Radiation toxicity; Hypofractionation; Margin reduction
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: The prospective pilot study will consist of two cohorts of patients: one cohort planned with the current standard PTV margin and the second cohort planned with the reduced margin validated from the retrospective study. The first cohort will be recruited while the retrospective study is being carried out and the second cohort will be accrued once the retrospective validation is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard margin (Active Comparator): Patient cohort planned with the current standard PTV margin
  Interventions: Radiation: External beam radiation therapy
- Reduced margin (Experimental): Patient cohort planned with the reduced margin validated from the retrospective study
  Interventions: Radiation: External beam radiation therapy

INTERVENTIONS:
Radiation: External beam radiation therapy — Patient will receive 60Gy in 20 fractions as per standard practice

SUMMARY:
The objectives of this study are:

1. Retrospectively validate a reduced margin schema for intermediate risk prostate hypofractionated VMAT treatments
2. Demonstrate in a prospective pilot clinical trial that patients planned and treated with the reduced margin schema will have reduced acute rectal toxicity

DETAILED DESCRIPTION:
Hypofractionated radiotherapy is being adopted as standard practice for intermediate risk prostate cancer patients. The objective of this project is to retrospectively validate whether reducing the Planning Target Volume (PTV), a margin placed around the prostate to account for movement and variability in patient placement, will have reduced acute rectal toxicity. The project will focus on patients with intermediate risk prostate cancer treated with hypofractionated Volumetric Modulated Arc Therapy (VMAT) from multiple institutions. The investigators intend to prospectively demonstrate that patients planned and treated with the reduced margin, along with using advanced image-guidance and consistent bladder and rectum preparation will have reduced acute rectal toxicity.

The project consists of two phases: phase one is a retrospective planning study and phase two is a prospective pilot clinical trial.

Phase one aims to validate the benefits of the proposed decrease in PTV margin by assessing whether the investigators can continue to deliver the intended radiation dose to the prostate while further sparing the rectum. This will be accomplished by evaluating the daily delivered dose on Cone-Beam Computed Tomography (CBCT), a daily scan performed during treatment that determines the location of the prostate and rectum. Using these CBCT scans, the investigators can reconstruct the radiation dose delivered to any organs of interest which was affected by their relative positions each day. There are two parts in this phase one retrospective planning study. Part one will focus on 30 intermediate risk prostate cancer cases already treated with hypofractionation (60 Gy in 20 fractions) using the standard PTV margins from all three participating institutions. All 30 cases will then be re-planned using the reduced PTV margin and dose reconstruction will be performed on daily CBCT to confirm adequate target coverage of the prostate. Part two aims to demonstrate that the reduced PTV margin can help enable hypofractionation. Thirty cases that were originally intended to receive a hypofractionated regimen of 60 Gy in 20 fractions but had to either switch to a standard fractionation treatment of 78 Gy in 39 fractions (a regimen used when 60Gy in 20 fractions is not achievable), or where there had to be compromised target coverage of the prostate, due to Organs at Risk (OAR) receiving unacceptable doses of radiation, will be selected. These cases will be re-planned with the validated smaller PTV margin to illustrate that they would now be eligible to receive hypofractionation due to the reduced dose to OARs.

Phase two aims to demonstrate that patients treated with the reduced PTV margin will have reduced acute rectal toxicity as evaluated by the Cancer Care Ontario (CCO) Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) Quality of Life (QOL) questionnaire. Two groups of patients will be accrued: one group of 25 patients will be planned and treated with the current standard PTV margin as the control group, while the second group of 25 patients will be planned and treated with the reduced PTV margin validated from the phase one retrospective study. A comparison of rectal toxicity scores between these two groups will then be carried out using the EPIC-CP questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with intermediate-risk prostate cancer receiving external beam radiotherapy
2. Age greater than or equal to 18 years
3. Agreeable to proposed follow-up schedule and able to complete quality of life questionnaire as proposed

Exclusion Criteria:

1. Previous radiotherapy to the pelvic region
2. Inflammatory bowel disease or chronic colitis.
3. Connective tissue disorders such as scleroderma.
4. Patients with hip replacements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patient diagnosed with intermediate-risk prostate cancer
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduced acute rectal toxicity from reduced PTV margin | 6 months
  Patients planned and treated with reduced PTV margin will have a change of 2 points in Cancer Care Ontario (CCO) Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) bowel symptom scores, demonstrating better toxicity outcomes. This patient reported outcome questionnaire evaluates bowel symptom scores in four aspects: rectal pain or urgency of bowel movement, increased frequency of bowel movements, overall problems with bowel movements, and bloody stools. Each aspect has a score ranging from 0 to 4. The total scores for an individual patient ranges from 0 to 16, with lower score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Beibei Zhang, PhD, Principal Investigator — Southlake Regional Health Centre
Locations (3):
- Canada (3):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Comprehensive Cancer Network: Prostate cancer, 2016. https://www.nccn.org/professionals/physician_gls/pdf/prostate.pdf
- [Background] Wortel RC, Incrocci L, Pos FJ, van der Heide UA, Lebesque JV, Aluwini S, Witte MG, Heemsbergen WD. Late Side Effects After Image Guided Intensity Modulated Radiation Therapy Compared to 3D-Conformal Radiation Therapy for Prostate Cancer: Results From 2 Prospective Cohorts. Int J Radiat Oncol Biol Phys. 2016 Jun 1;95(2):680-9. doi: 10.1016/j.ijrobp.2016.01.031. Epub 2016 Jan 22. PMID 27055398
- [Background] Dearnaley DP, Khoo VS, Norman AR, Meyer L, Nahum A, Tait D, Yarnold J, Horwich A. Comparison of radiation side-effects of conformal and conventional radiotherapy in prostate cancer: a randomised trial. Lancet. 1999 Jan 23;353(9149):267-72. doi: 10.1016/S0140-6736(98)05180-0. PMID 9929018
- [Background] Alayed Y et al: Clinical impact of reducing planning target volume margins during radiation therapy for localized prostate cancer: early outcomes of a 2-stage prospective trial. Int J Radiat Oncol Biol Phys 93:(S)E249, 2015
- [Background] Nijkamp J, Pos FJ, Nuver TT, de Jong R, Remeijer P, Sonke JJ, Lebesque JV. Adaptive radiotherapy for prostate cancer using kilovoltage cone-beam computed tomography: first clinical results. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):75-82. doi: 10.1016/j.ijrobp.2007.05.046. Epub 2007 Sep 17. PMID 17869445
- [Background] Gill SK, Reddy K, Campbell N, Chen C, Pearson D. Determination of optimal PTV margin for patients receiving CBCT-guided prostate IMRT: comparative analysis based on CBCT dose calculation with four different margins. J Appl Clin Med Phys. 2015 Nov 8;16(6):252-262. doi: 10.1120/jacmp.v16i6.5691. PMID 26699581
- [Background] Battista JJ, Johnson C, Turnbull D, Kempe J, Bzdusek K, Van Dyk J, Bauman G. Dosimetric and radiobiological consequences of computed tomography-guided adaptive strategies for intensity modulated radiation therapy of the prostate. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):874-80. doi: 10.1016/j.ijrobp.2013.07.006. Epub 2013 Aug 24. PMID 23978708
- [Background] Nuver TT, Hoogeman MS, Remeijer P, van Herk M, Lebesque JV. An adaptive off-line procedure for radiotherapy of prostate cancer. Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1559-67. doi: 10.1016/j.ijrobp.2006.12.010. Epub 2007 Feb 15. PMID 17306934
- [Background] Engels B, Soete G, Gevaert T, Storme G, Michielsen D, De Ridder M. Impact of planning target volume margins and rectal distention on biochemical failure in image-guided radiotherapy of prostate cancer. Radiother Oncol. 2014 Apr;111(1):106-9. doi: 10.1016/j.radonc.2014.02.009. Epub 2014 Mar 13. PMID 24631146
- [Background] Quon HC et al: PATRIOT trial: randomized phase II study of prostate stereotactic body radiotherapy comparing 11 versus 29 days overall treatment time. J Clin Oncol 33:(S)6-6, 2015.
- [Background] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Background] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- [Background] Chang P, Szymanski KM, Dunn RL, Chipman JJ, Litwin MS, Nguyen PL, Sweeney CJ, Cook R, Wagner AA, DeWolf WC, Bubley GJ, Funches R, Aronovitz JA, Wei JT, Sanda MG. Expanded prostate cancer index composite for clinical practice: development and validation of a practical health related quality of life instrument for use in the routine clinical care of patients with prostate cancer. J Urol. 2011 Sep;186(3):865-72. doi: 10.1016/j.juro.2011.04.085. Epub 2011 Jul 23. PMID 21788038
- [Background] Howell D et al: Feasibility of implementing EPIC-CP: recommendations to enhance the quality of person-centred clinical care of men with early-stage prostate cancer. Cancer Care Ontario report.
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Korzeniowski M, Kalyvas M, Mahmud A, Shenfield C, Tong C, Zaza K, Howell D, Brundage M. Piloting prostate cancer patient-reported outcomesin clinical practice. Support Care Cancer. 2016 May;24(5):1983-1990. doi: 10.1007/s00520-015-2949-5. Epub 2015 Oct 24. PMID 26498748
- [Background] Lee WR et al: RTOG 0415: A phase III randomized study of hypofractionated 3DCRT/IMRT versus conventionally fractionated 3DCRT/IMRT in patients treated for favorable-risk prostate cancer.